CLINICAL TRIAL: NCT04189315
Title: A Phase 4, Randomized, Multicenter, Open-Label, 2-Dosage Regimen, Safety and Tolerability, Efficacy, Pharmacokinetic, and Pharmacodynamic Study of Asfotase Alfa in Adult Patients With Pediatric-Onset Hypophosphatasia
Brief Title: Relieving Burden of Hypophosphatasia in Adults With Functional Impairment Due to Chronic Disease
Acronym: REBUILD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: R&D portfolio review and in light of the global impact of the COVID-19 pandemic
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA-HPP-406
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; HPP; Pediatric-Onset; Asfotase Alfa
MeSH Terms: conditions — Hypophosphatasia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 Asfotase Alfa (Experimental): Participants will be administered asfotase alfa per approved dose for 36 weeks.
  Interventions: Drug: asfotase alfa
- Group 2 Asfotase Alfa (Experimental): Participants will be administered asfotase alfa per approved dose for 12 weeks and then asfotase alfa at a lower dose for 24 weeks.
  Interventions: Drug: asfotase alfa

INTERVENTIONS:
Drug: asfotase alfa — Asfotase alfa is administered subcutaneously.

SUMMARY:
The study will evaluate safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of 2 different doses (approved dose and lower dose) of asfotase alfa in adult participants with pediatric-onset hypophosphatasia (HPP).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years at the time of signing the informed consent form
* Clinical diagnosis of pediatric-onset HPP based on signs and symptoms consistent with HPP
* Past medical history that includes at least one nonvertebral fracture (or pseudofracture) incurred without evidence of significant trauma.
* The presence of a current fracture is not necessary, but for participants with current unhealed fracture(s) or pseudofracture(s) of the lower extremity(ies) (that is, femoral, tibial, fibular, metatarsal) documentation must be provided of the presence of these fractures for at least 3 months prior to screening (with or without surgical intervention)

Exclusion Criteria:

* Medical condition, serious concurrent or recurrent illness and/or injury, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance or the assessment of study endpoints, including all protocol required evaluations and follow up activities, or may put the patient at risk
* Primary or secondary hyperparathyroidism or hypoparathyroidism
* History of hypersensitivity to any ingredient contained in asfotase alfa
* Oral bisphosphonate use within 6 to 12 months (depending on the half-life of the drug as assessed by the investigator) and intravenous (IV) bisphosphonate use within 12 months prior to screening
* Denosumab use within 18 months prior to screening
* Asfotase alfa use within 6 months prior to screening
* Teriparatide/parathyroid hormone analog use within 2 months prior to screening
* Treatment with strontium or sclerostin inhibitors within 6 months prior to the first dose of study drug
* Vitamin B6 use for at least 2 weeks prior to screening
* Serum 25-hydroxy (25-OH) vitamin D below 20 nanogram (ng)/milliliter (mL), with repletion and recheck allowed at screening (results from local laboratory may be used if within 4 weeks of screening)
* Female patients who are pregnant, planning to become pregnant, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline To Week 36 In Plasma Concentrations Of Inorganic Pyrophosphate (PPi) In Group 1 | Baseline, Week 36

SECONDARY OUTCOMES:
Change From Baseline To Week 36 In Plasma Concentrations Of PPi In Group 2 | Baseline, Week 36
Change From Baseline To Week 36 In The 36-item Short-Form Survey (SF-36) Physical Component Summary (PCS) Score In Groups 1 And 2 | Baseline, Week 36
Change From Baseline To Week 36 In The Repeated Chair Stand Test (A Component Of The Short Physical Performance Battery [SPPB]) In Groups 1 And 2 | Baseline, Week 36

IPD SHARING:
Plan to Share IPD: No